CLINICAL TRIAL: NCT05568992
Title: Prospective, Randomized Controlled Study to Evaluate the Effect of Artificial Intelligence Assisted Optical Diagnosis of Advanced Adenomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Renji KY[2019]009
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Advanced Adenoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI assisted group (Experimental): AI assisted endoscopist' optical detection of advanced adenomas among 100 images of polyps
  Interventions: Device: AI system of optical detection of advanced adenomas
- non-AI assisted group (No Intervention): Endoscopist' optical detection of advanced adenomas among 100 images of polyps using their experience of colonoscopy

INTERVENTIONS:
Device: AI system of optical detection of advanced adenomas — AI system of optical detection of advanced adenomas
  Arms: AI assisted group

SUMMARY:
This study is a clinical validation of our developed a computer-aided optical dignosis of advanced adenoma using non-magnified NBI image. This study is a randomized clinical trial comparing endoscopists' optical recognition of advanced adenoma for sending to histological examination with our computer-aided system. The hypothesis of the study is that the developed computer-aided system increases the percent of sending actual advanced adenoma Intelligence Assisted Optical Diagnosis of Advanced Adenomas

DETAILED DESCRIPTION:
Colorectal polyp diagnosis is based on endoscopic resection and histological analysis. An accurate optical diagnosis could avoid histological lesion of smaller lesions, reducing the costs associated with histological diagnosis. However, it should be noted this policy could only be applied in diminutive polys considering high proposition of advanced adenomas in polyps more than 5 mm. In addition, optical diagnosis criteria of advanced adenomas have not been validated for finding advanced adenomas among adenoma polyps. If as many as advanced adenomas as possible could be differentiated from non-advanced adenomas and be further sent for histological examination, this policy could be generalized to small polyps.

Considering this situation, the investigators tried to develop computer-aided optical dignosis of advanced adenoma using non-magnified NBI image with preliminary, satisfied results. In this study, the investigators next validate the investigators' developed computer-aided system for detecting advanced adenomas by comparing endoscopists' optical detection of advanced adenomas with or without the investigators' computer-aided system.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists with NBI experience

Exclusion Criteria:

* Endoscopists without colonoscopy and NBI experience

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Proportion of advanced adenomas for sending to histological examination | 1 day
  Proportion of advanced adenomas for sending to histological examination

SECONDARY OUTCOMES:
Optical diagnostic accuracy of non-advanced adenomas under high confidence | 1 day
  Optical diagnostic accuracy of non-advanced adenomas under high confidence
Proportion of high confidence optical diagnosis of polyps | 1 day
  Proportion of high confidence optical diagnosis of polyps

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No